CLINICAL TRIAL: NCT04107948
Title: Efficiency of an Optimized Care Organization for Fibromyalgia Patients Within the Group of Hospitals of Loire Territory. Interventional Study Aimed at Changing Behaviour in Terms of Physical Activity and Sedentary
Brief Title: Efficiency of an Optimized Care Organization for Fibromyalgia Patients. The FIMOUV 2 Study
Acronym: FIMOUV 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18PH223; 2019-A02221-56 (Other: ANSM)
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia; Physical Activity
Keywords: sedentary time; therapeutic education sessions
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Sedentary Behavior | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fibromyalgia patients with physical activity program (Experimental): Two weekly exercise sessions at the university hospital of St-Etienne for 1 month then relay outside in a sports association or club certified "Sports Health" in the Loire (42) or Haute-Loire (43) for 2 months.
  Interventions: Other: physical activity program
- fibromyalgia patients with physical activity at home (Other): Advice and recommendations of physical activity at home (= current clinical practice, from 1 to 3 sessions per week in autonomy).
  Interventions: Other: Advice and recommendations of physical activity at home

INTERVENTIONS:
Other: physical activity program — Two weekly exercise sessions at the university hospital of St-Etienne for 1 month then relay outside in a sports association or club certified "Sports Health" in the Loire (42), Haute-Loire (43) or Ardèche (07) for 2 months.
  Arms: fibromyalgia patients with physical activity program
Other: Advice and recommendations of physical activity at home — Advice and recommendations of physical activity at home (= current clinical practice, from 1 to 3 sessions per week in autonomy).
  Arms: fibromyalgia patients with physical activity at home

SUMMARY:
Fibromyalgia affects 2 to 5% of adults in the general population. Patients describe a combination of symptoms centred around fatigue not induced by exercise and not relieved by rest.

The diagnosis of fibromyalgia is self-perpetuating by the deconditioning, consequence of a reduced muscle mass due to inactivity and periods of prolonged rest.

Thus, it seems fundamental to develop other non-drug approaches: among them, adapted physical activity is recommended by most learned societies because of a good level of evidence (Level 1, Grade A). The question remains, however, whether simple advice to resume physical activity is sufficient (routine care with medical assessment at 3 months) or whether a physical activity supervised inside and outside the hospital is not more relevant.

DETAILED DESCRIPTION:
In order to set up an optimal patient path within the Group of hospitals of Loire territory, the working group composed of doctors from different specialities of the department considered it important to carry out a randomised study evaluating the effectiveness of a healthcare organisation combining:

* an adapted and supervised physical activity intervention (1 month hospital initiation then 2 months in town)
* therapeutic education sessions for the patient with motivational interviews Compared to usual clinical practice (adapted physical activity adapted in autonomy at home + therapeutic patient education sessions with motivational interviews).

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with fibromyalgia according to ACR (American College of rheumatology) criteria (total score WPI (Widespread Pain Index) + SS (Severity Scale) ) ≥ 13
* French writing and speaking
* Sedentary or low level of activity (less than 150 minutes of regular physical activity per week at the time of inclusion)
* Signature of informed consent

Exclusion Criteria:

* Cardiac or respiratory diseases that contraindicate the practice of physical activity
* Significant co-morbidities that contraindicate the practice of physical activity: associated cardiac pathologies (severe rhythm disorders such as rapid atrial fibrillation), respiratory pathologies (severe obstructive or severe respiratory insufficiency), disabling joint pathologies (knee osteoarthritis or osteoarthritis of the hip) training on a treadmill or on a high intensity bike).
* Impossibility of submitting to the medical monitoring of the program for geographical, social or psychological reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
physical activity | 12 months
  Measure the durability of adherence/therapeutic compliance of fibromyalgia patients based on an objective measurement of physical activity: average measured from 7 days of actimetry, Actigraph

SECONDARY OUTCOMES:
sedentary | 12 and 24 months
  Measure the durability of adhesion/therapeutic compliance of fibromyalgia patients based on an objective measurement of sedentary : average measured from 7 days of actimetry, Actigraph
physical activity | 0, 1, 3, 6, 12 and 24 months
  Objective and repeated measurement of physical activity over 7 days using actimetry, Actigraph
sedentary | 0, 1, 3, 6, 12 and 24 months
  Objective and repeated measurement of sedentary over 7 days using actimetry, Actigraph
health status | 0, 1, 3, 6, 12 and 24 months
  measured with Patient Global Impression of Change (PGIC) : on a 7-point scale, rated from 1 for "much worse" to 7 for "much better". It is a simple and practical evaluation tool to use. The combination of the level of achievement via the Patient Global Impression of Change and the initial documentation of the patient's objectives via the shared educational assessment is a relevant and understandable approach for the patient.
fatigue | 0, 1, 3, 6, 12 and 24 months
  assessed by Fatigue Severity Scale. This is a short questionnaire of 9 questions to which the patient answers on a scale from 1 to 7.
  Simply add the scores and divide by 9 - you get a result on 7 points. The higher the result, the greater the fatigue. Several studies speak of a threshold at 5.5
Quality of sleep | 0, 1, 3, 6, 12 and 24 months
  assessed by the Pittsburgh. The questionnaire includes 19 self-assessment questions and 5 questions for the spouse or roommate (if any). Only self-assessment questions are included in the score.
  The 19 self-assessment questions combine to give 7 components" of the score with each component receiving a score of 0 to 3.
  In all cases, a score of 0 indicates that there is no difficulty while a score of 3 indicates the existence of severe difficulties. The 7 components of the score add up to give an overall score from 0 to 21 points, 0 meaning that there is no difficulty, and 21 indicating on the contrary major difficulties.
Anxiety and Depression | 0, 1, 3, 6, 12 and 24 months
  assessed by the Hospital Anxiety and Depression Scale (HADS) : An overall score of 19 or more indicates a major depressive episode. An overall score of 13 corresponds to adjustment disorders and minor depression.
pain catastrophizing | 0, 1, 3, 6, 12 and 24 months
  assessed by the PCS (pain catastrophizing scale) assessing catastrophism : there are thirteen statements describing different thoughts and emotions that may be associated with pain. the person must indicate how painful these thoughts and emotions are. From 0= not at all to 4 = all the time
pain evaluation | 6 and 12 months
  assessed by analog visual evaluation of pain (0= no pain and 10 = very painful)
fatigue evaluation | 6 and 12 months
  assessed by analog visual evaluation of fatigue (0= no fatigue and 10 = maximum fatigue)
muscle power | 0, 1 and 3 months
  evaluated by dynamometry on a stress platform (arms and legs) and by a pocket dynamometer.
muscular endurance | 0, 1 and 3 months
  evaluated by dynamometry on a stress platform (arms and legs).
gas exchange measurement | 0, 1 and 3 months
  evaluated during a stress test
fatigue | 0, 1 and 3 months
  evaluated with Baroreflex Sensitivity. measurement of the slope of the baroreflex
quantification of physical activity in meter-h/week | 0, 1, 3, 6,12 and 24 months
  evaluated by the APAQ : Adult Physical Activity Questionnaire
sedentary times in hours/day | 0, 1, 3, 6, 12 and 24 months
  evaluated by the APAQ : Adult Physical Activity Questionnaire
patient adherence | 6 and 12 months
  number of sessions performed
Direct medical costs | 12 months
  consultations, examinations, hospitalizations in euros
Direct non-medical costs | 12 and 24 months
  transport
Cost of lost productivity | 12 and 24 months
  time not worked

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, Principal Investigator — CHU de Saint Etienne
Locations (7):
- France (7):
  - CH d'ANNONAY, Annonay
  - CH de Firminy, Firminy
  - CH de MONTBRISON, Montbrison
  - CH de Rive de Gier, Rive-de-Gier
  - CH de ROANNE, Roanne
  - CH du Gier, Saint-Chamond
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colas C, Jumel A, Vericel MP, Barth N, Manzanares J, Goutte J, Fontana L, Feasson L, Hupin D, Guyot J. Understanding Experiences of Fibromyalgia Patients Involved in the Fimouv Study During COVID-19 Lockdown. Front Psychol. 2021 Jul 20;12:645092. doi: 10.3389/fpsyg.2021.645092. eCollection 2021. PMID 34354626
- [Derived] Colas C, Goutte J, Creac'h C, Fontana L, Vericel MP, Manzanares J, Peuriere M, Akrour M, Martin C, Presles E, Barth N, Guyot J, Garros M, Trombert B, Massoubre C, Roche F, Feasson L, Marotte H, Cathebras P, Hupin D. Efficiency of an Optimized Care Organization in Fibromyalgia Patients: The From Intent to Move (FIMOUV) Study Protocol of a Randomized Controlled Trial. Front Public Health. 2021 May 25;9:554291. doi: 10.3389/fpubh.2021.554291. eCollection 2021. PMID 34113593